CLINICAL TRIAL: NCT04022811
Title: Bromfenac Ophthalmic Solution 0.1% for Postoperative Ocular Pain and Inflammation Related To Pterygium Surgery
Brief Title: Effect of Bromfenac on Pain Related to Pterygium Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018KYPJ101
Record Dates: First submitted 2018-05-22; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Pterygium; Pain
Keywords: Pterygium; Bromofenac; Pain
MeSH Terms: conditions — Pterygium; Pain | interventions — bromfenac; Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Artificial tears (Experimental): 0.1% bromfenac VS Artificial tears
  Interventions: Drug: 0.1% bromfenac

INTERVENTIONS:
Drug: 0.1% bromfenac — the patients received the use of the Ponacore 3 days before and 7 days after the operation. Local eye drops, 2 times a day.
  Other Names: 0.5%Tobramycin dexamethasone; 0.3% sodium hyaluronate

SUMMARY:
To evaluate the efficacy and ocular safety of bromfenac ophthalmic solution (bromfenac) 0.1% dosed twice daily for the treatment of ocular inflammation and pain after pterygium excision with amniotic membrane transplantation(AMT).

DETAILED DESCRIPTION:
Patients scheduled to undergo pterygium excision with AMT were randomized to receive added topical bromfenac or artificial lacrima at 3 days before and 7 days after the surgery. Pain intensity was evaluated with the visual analog scale(VAS) and present pain index(PPI) with the short form of the McGill Pain Questionnaire. psychological state used Self-rating of Depression Scale(SDS) and Self-rating of Anxiety Scale (SAS) to assess. Ocular inflammation was assessed with an automated bulbar redness grading technique. The irritative symptoms evaluation was carried out by an independent investigator at each visit with questionnaires of ocular symptom scores(OSS). Corneal epithelial healing rate was calculated after following up. All patients had follow-ups at the day 1, day 3, day7 and day 10.

ELIGIBILITY:
Inclusion criteria

1. Patients with unilateral or double pterygium
2. The gender is not limited, age 45-75 years old
3. intraocular pressure <21mmHg
4. follow the preoperative and postoperative drug regimen and ensure regular follow-up

Exclusion Criteria

1. Patient factors: lack of cooperation and poor compliance.
2. Severe dry eye, Sjogren's syndrome, cicatricial pemphigoid, and other systemic diseases that seriously affect the structure or function of the ocular surface.
3. Glaucoma or high intraocular pressure (above 21 mmHg), active uveitis, retinal detachment and other diseases.
4. History of systemic diseases, such as uncontrolled diabetes and hypertension, rosacea, severely impaired cardiopulmonary function or other diseases that cannot tolerate surgery; central nervous system disorders affect patient perception, trigeminal neuritis, trigeminal neuralgia, and tongue Pharyngeal neuralgia, migraine and period of toothache attack.
5. history of drug allergies, such as NSAID drugs, tobramycin, anesthetics and so on. Smokers and alcoholics (smoking volume >15 cigarettes/day, pure alcohol consumption>100 ml/week).
6. Other history of eye surgery, such as history of eye trauma, history of glaucoma surgery, history of cataract surgery, history of retinal surgery, or other serious injuries to the eyelids, conjunctiva, cornea, and other tissues of the eye surface.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
visual analog scale(VAS) | Change from Baseline VAS at 10 days
  The VAS pain score provides an intensity score of the pain experienced. The VAS allows the patient to self-rate his or her pain on a 0 to 10 horizontal grading scale of subjective pain assessment with 0 as "no pain at all" and 10 being "the most severe intolerable pain I have ever experienced."
present pain intensity index(PPI) | Change from Baseline PPI at 10 days
  The PPI scale is a measure of the magnitude of pain experienced by an individual and is a six-point verbal rating scale that indicates overall pain intensity and includes six levels (0, none; 1, mild; 2, discomforting; 3, distressing; 4, horrible; and 5, excruciating). Higher numbers indicate more severe pain.

SECONDARY OUTCOMES:
corneal epithelium healing(CEH) | Change from Baseline corneal epithelial defect at 10 days
  Took the anterior segment photography and slit lamp examination parallel sodium fluorescein staining. The corneal epithelial defect area was stained with fluorescein sodium. Corneal epithelial healing rate is obtained by calculating the difference of the corneal epithelial defect area on day1 from day10, then divided by days.
Inflammation Evaluation by temporal conjunctival hyperaemia index (TCHI) | Change from Baseline TCHI at 10 days
  Ocular inflammation was assessed with an automated bulbar redness grading technique, the Oculus Keratograph○R5M (Oculus Optikgerate GmbH, Wetzlar, Germany) by temporal conjunctival hyperaemia index (TCHI). The Oculus Keratograph 5M returns redness using a clinical grading scale of 0.0-4.0 in 0.1 steps.we choose TCHI to evaluate the degree of ocular inflammation, which the grade of 1.2 or less is considered a physiologic degree of bulbar redness.
Symptoms Evaluation by ocular symptom scores(OSS) | Change from Baseline OSS at 10 days
  The irritative symptoms evaluation by ocular symptom scores(OSS),which was carried out by an independent investigator at each visit with questionnaires of ocular symptom scores(OSS), which included grading of their symptoms (pain, foreign body sensation, burning sensation, visual fatigue and dryness) using a 4-point scale. The patients determine the quality of irritative symptom by selecting one of the options: None = 0, Perceptible or intermittent fatigue=1, Obvious visual fatigue but tolerable=2, Apparent visual fatigue and hard to bear=3. Higher numbers indicate more severe irritative symptom.
psychological state changes of depression was evaluated with Self-rating Depression Scale(SDS) | Change from Baseline SDS at 10 days
  In the main component of the SDS , patients are asked 20 questions about Mental and physical feelings of emotional experience, and the patients determine the quality of emotion by selecting one of the options: Occasionally=1, sometimes=2, often=3, and continuously=4. 10 questions are scored forward, the other 10 questions are scored backward. The total score is multiplied by an integer of 1.25 to get the standard score. According to Chinese norms, the cut-off value of SDS standard score is 53, 53-62 is mild, 63-72 is moderate, over 72 is severe, and lower than 53 belongs to the normal.
psychological state changes of anxiety was evaluated with Self-rating Anxiety Scale(SAS) | Change from Baseline SAS at 10 days
  In the main component of the SAS , patients are asked 20 questions about Mental and physical feelings of emotional experience, and the patients determine the quality of emotion by selecting one of the options: Occasionally=1, sometimes=2, often=3, and continuously=4. 10 questions are scored forward, the other 10 questions are scored backward. The total score is multiplied by an integer of 1.25 to get the standard score. According to Chinese norms, the cut-off value of SAS standard score is 53, 53-62 is mild, 63-72 is moderate, over 72 is severe, and lower than 53 belongs to the normal.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, DOC, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (2):
- China (2):
  - Zhongshan Opthalmic Center, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walters TR, Goldberg DF, Peace JH, Gow JA; Bromfenac Ophthalmic Solution 0.07% Once Daily Study Group. Bromfenac ophthalmic solution 0.07% dosed once daily for cataract surgery: results of 2 randomized controlled trials. Ophthalmology. 2014 Jan;121(1):25-33. doi: 10.1016/j.ophtha.2013.07.006. Epub 2013 Sep 8. PMID 24021896
- [Background] Rajpal RK, Ross B, Rajpal SD, Hoang K. Bromfenac ophthalmic solution for the treatment of postoperative ocular pain and inflammation: safety, efficacy, and patient adherence. Patient Prefer Adherence. 2014 Jun 25;8:925-31. doi: 10.2147/PPA.S46667. eCollection 2014. PMID 25028541
- [Background] Hoy SM. Bromfenac Ophthalmic Solution 0.07%: A Review of Its Use After Cataract Surgery. Clin Drug Investig. 2015 Aug;35(8):525-9. doi: 10.1007/s40261-015-0309-3. PMID 26177719
- [Background] Donnenfeld ED, Holland EJ, Stewart RH, Gow JA, Grillone LR; Bromfenac Ophthalmic Solution 0.09% (Xibrom) Study Group. Bromfenac ophthalmic solution 0.09% (Xibrom) for postoperative ocular pain and inflammation. Ophthalmology. 2007 Sep;114(9):1653-62. doi: 10.1016/j.ophtha.2006.12.029. Epub 2007 Apr 19. PMID 17445902
- [Background] Henderson BA, Gayton JL, Chandler SP, Gow JA, Klier SM, McNamara TR; Bromfenac Ophthalmic Solution (Bromday) Once Daily Study Group. Safety and efficacy of bromfenac ophthalmic solution (Bromday) dosed once daily for postoperative ocular inflammation and pain. Ophthalmology. 2011 Nov;118(11):2120-7. doi: 10.1016/j.ophtha.2011.04.035. Epub 2011 Jul 16. PMID 21762992
- [Background] Silverstein SM, Cable MG, Sadri E, Peace JH, Fong R, Chandler SP, Gow JA, Klier SM, McNamara TR; Bromfenac Ophthalmic Solution Once Daily (Bromday) Study Group. Once daily dosing of bromfenac ophthalmic solution 0.09% for postoperative ocular inflammation and pain. Curr Med Res Opin. 2011 Sep;27(9):1693-703. doi: 10.1185/03007995.2011.597663. Epub 2011 Jul 14. PMID 21751945